CLINICAL TRIAL: NCT04117139
Title: The Diagnostic Value of 18F-2-fluoro-2-deoxy-D-glucose Fluorodeoxyglucose-Positron-Emission-Tomography/Magnetic-Resonance Imaging (PET/MRI) for Cervical Lymph Node Metastasis in Head and Neck Squamous Cell Carcinoma
Brief Title: The Diagnostic Value of PET/MRI in Head and Neck Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Odense University Hospital (Other)
Collaborators: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Chadi Nimeh Abdel-Halim, Medical Doctor and Principal Investigator, Odense University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HNC PET/MRI
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Lymph Node Metastases
Keywords: Positron-Emission-Tomography/Magnetic Resonance Imaging; PET/MRI; Cancer staging
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Lymphatic Metastasis | interventions — Positron-Emission Tomography; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Group (Other): In addition to other standard imaging modalities in the fast track cancer program, included patients will have a PET/MRI done.
  Interventions: Diagnostic Test: PET/MRI

INTERVENTIONS:
Diagnostic Test: PET/MRI — A PET/MRI of the Head and Neck region is done for all patients included in the project.
  Other Names: 18F-FDG-PET/MRI; FDG-PET/MRI; PET/MR; PET-MR; Positron-Emission-Tomography/Magnetic Resonance Imaging

SUMMARY:
This study investigates the diagnostic value of PET/MRI for cervical lymph node metastases from head and neck squamous cell carcinomas.

DETAILED DESCRIPTION:
The Danish fast-track cancer program standardizes the work-up of patients suspected of head and neck cancer. Currently, the guidelines recommend head and neck magnetic resonance imaging (MRI) as the standard imaging modality for assessment of the primary tumor site and potential nodal metastases. However, recent studies have shown advantages in the use of 18F-FDG-PET (PET) combined with computed tomography (CT) due to its superiority in detecting metastases and synchronous cancers.

During the last couple of years PET/MRI has been introduced. MRI is known to provide the highest anatomic detail in the head and neck region, and preliminary studies show promising results. However, the evidence is still very sparse.

The purpose of the project is to investigate the diagnostic value of PET/MRI in patients with head and neck squamous cell carcinoma. The hypothesis is that PET/MRI provides a more precise diagnosis of regional lymph node metastases, and thus, make the surgical treatment of the neck more accurate and less invasive resulting in reduced morbidity.

The project is designed as a prospective cohort study based on paired data with head-to-head comparison of CT, MRI, PET/CT and PET/MRI. Patients will be included from the head and neck cancer fast-track program at the Center of Head and Neck Cancer, Odense University Hospital (OUH).

Included patients will be offered PET/MRI in addition to the conventional fast-track imaging. The description of the images will be made blinded. When a neck dissection of the lymph nodes is made, the lymph nodes will be separated in defined regions. The diagnostic accuracy of the individual imaging modalities is assessed for each neck level with histology as standard reference.

ELIGIBILITY:
Inclusion Criteria:

Patients either suspected of or with histologically verified:

* Relapse of head and neck squamous cell cancer with involvement of regional lymph node(s)
* Cervical lymph node metastasis with unknown primary tumor site
* Oral cavity squamous cell carcinoma
* Oropharyngeal squamous cell cancer planned for trans oral robotic surgery

Exclusion Criteria:

* Patients who cannot have a PET/MRI performed for different reasons (allergy, claustrophobia, medical implants)
* Patients who had surgery, infection or other inflammatory inducing conditions on the neck within the last 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of PET/MRI for Malignancy in Regional Lymph Nodes | 7-10 days
  PET/MRI scans are compared to histology as the golden standard to determine the diagnostic accuracy of PET/MRI for malignancy in regional lymph nodes

SECONDARY OUTCOMES:
Diagnostic Accuracy of PET/MRI for Extracapsular Lymph Node Spread | 7-10 days
  PET/MRI scans are compared to histology as the golden standard to determine the diagnostic accuracy of PET/MRI for extracapsular spread in regional lymph nodes

CONTACTS AND LOCATIONS:
Overall Officials: Chadi N. Abdel-Halim, M.D., Principal Investigator — Odense University Hospital
Locations (1):
- Department of ORL - Head & Neck Surgery and Audiology, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No